CLINICAL TRIAL: NCT06753526
Title: L-Arginine Role for Stone Lower Ureter : A Randomized Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Mohammed Ahmed Elsherief, lecturer of urology at faculty of medicine ,sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-05-09PD
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-05

CONDITIONS: Stone Lower Ureter
Keywords: stone; medical expulsive therapy
MeSH Terms: conditions — Calculi | interventions — Anti-Inflammatory Agents, Non-Steroidal; Arginine; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (Placebo Comparator): about 53 patient, received NSAIDs
  Interventions: Drug: NSAID
- Group II (Active Comparator): about 53 patients received L-arginine 1000 mg once daily
  Interventions: Drug: L-Arginine, 500 Mg Oral Capsule
- group III (Active Comparator): included 51 patients who received Tamsulosin 0.4 mg once daily.
  Interventions: Drug: Tamsulosin 0.4 mg QD

INTERVENTIONS:
Drug: NSAID — For 1st group of patients
  Arms: Group I
Drug: L-Arginine, 500 Mg Oral Capsule — group 2by twice dose
  Arms: Group II
Drug: Tamsulosin 0.4 mg QD — group 3 by once per day
  Arms: group III

SUMMARY:
To evaluate the effects of L-Arginine 1000mg once daily as a medical expulsive therapy (MET) for lower ureter stones.

DETAILED DESCRIPTION:
Urolithiasis is a common disease worldwide and its incidence is growing [1]. Urinary stones are frequently located in the ureter and most ureteral stones are reported to be located distally [2]. Stones < 3 mm in diameter have a better chance to pass spontaneously in the majority of cases, whereas stones > 6 mm in the ureter are unlikely to pass in most situations [3].

Therefore, active watchful waiting forms one of the treatment options in some clinical scenarios.

Minimal invasive treatment strategies such as extracorporeal shockwave lithotripsy and ureteroscopy are frequently applied procedures in ureteral stone disease. However, indications for watchful waiting might be extended by the addition of so-called 'expulsive medical therapy'.

Nitric Oxide (NO) L -Arginine-derived NO is the major inhibitory NANC neurotransmitter in the lower urinary tract [4]. Neuronal NO synthase (NOS)-positive neuronal axons and nerve-ending-like structures have been detected in muscular layers of the human ureter suggesting that ureteral relaxation may involve the NO pathway [5]. NOS-reactive nerves have also been demonstrated immunohistochemically in the human intravesical ureter.

A recent study suggested that the L-arginine/NO/cyclic GMP pathway may play a role in the regulation of the valve function of the ureterovesical junction [6].

NO has been shown to have a smooth muscle-relaxing effect in various animal species and humans. Mastrangelo et al. [7] showed that urothelium-produced NO inhibits contractile responses in the proximal ureter in rats. NOS was also demonstrated in the nerve fibers of the porcine intravesical ureter and was suggested to mediate the inhibitory neurotransmission [8].

Neuronal NOS-positive nerves have been shown in the human ureter, particularly in the distal part which seems to have an important function regarding peristalsis and ureterovesical junction motility [9]. Therefore, this pathway may also be a new target for new drugs producing relaxation of the human ureter.

In renal colic The severe pain of renal colic (RC) caused by urinary stone disease has an occurrence rate of 1-10% for each person per their lives and accounts for 2% of all admittances to the emergency department [10-12]. The stone passing into the ureter produces high intraluminal pressure, which may cause contractions of the smooth muscles of the ureter and induce irritation and obstruction, which hereby produces spasms that lead to unbearable pain [13,14].

Nitric oxide (NO), which is synthesized from L-arginine, has a role in the physiopathology of RC. Because axons and neuronal endings that are positive for neuronal nitric oxide synthase (nNOS) reside in the human ureter, NOS, which participates in the synthesis of NO may be related to The hypothetical relationship between NO and RC is expressed in the hypothesis that NO can cause the progression of a stone to be easier and stiffer with a dilatation effect on the ureter where the smooth muscle is located. The possible relationship between RC and endothelial NOS (eNOS), which is a different isoenzyme that is involved in the synthesis of NO that functions in smooth muscle organs such as the ureter, has been left mostly unexplored to this day. Endothelial NOS, which is coded for by a gene that is located on the long arm of the 7th chromosome, has a role in the synthesis of NO, which relaxes the smooth muscles of the gastrointestinal and cardiovascular systems and acts in other pathophysiological processes [16,17].

Objectives To evaluate the effects of L-Arginine once daily as a medical expulsive therapy for stone lower ureter by conducting a randomized study Study Design The design of the research will be a prospective randomized controlled study. Study Setting/Location The study will be conducted in a single tertiary center at the Urology department in Sohag University, Egypt.

Local ethics committee approval was obtained for this trial. all participants will be discussed to participate in this study.

Patients and Methods Inclusion criteria All the participants, older than 18 years old ureter stones in size between 4 and 10 mm single stone Exclusion criteria Acute azotemia, stones larger than 8mm, solitary kidney, drainage due to urinary tract infection, symptomatic urinary system infection, impacted status, concomitant use of a-blockers, anticholinergics, corticosteroids, calcium channel blockers, and analgesics; severe hydronephrosis, multiple stones, pregnancy, previous ureter and bladder operations, anatomic urinary system abnormalities, benign prostate hyperplasia, uncontrolled hypertension (systolic blood pressure≥180 mmHg, diastolic blood pressure≥110 mmHg), bilateral ureter stone, stones bigger than 10 mm, residual stone after any procedure (shock wave lithotripsy, ureterolithotripsy, ureterolithotomy, etc.), Study procedure Evaluations included

1. Detailed history
2. Physical examination
3. Urinalysis & urine culture
4. Renal function tests
5. Ultrasonography
6. PUT
7. Computed tomography of the urinary tract. Intramural ureteral stones were diagnosed using kidney-ureter-bladder radiography and urinary system ultrasonography A computed tomography (CT) scan was performed on suspected patients

Recorded details included:

Baseline characteristics of patients.

* Number of patients
* age
* gender
* stone's laterality,
* stone's location
* stone's surface area (Stone size)
* degree of hydronephrosis medical history, family history, complaints secondary to pain and the presence of fever, blood pressure, cardiac pulse, and respiratory rate abnormalities of the RC. Follow up Patients will followed weekly for 4 weeks by ultrasonography and/or KUB Follow up details
* Spontaneous stone expulsion rates (SER),
* stone expulsion time,
* the number of daily colic episodes
* total required analgesic dosage of the patients

Study Procedures

Patients meeting the inclusion criteria will be randomly allocated to 3 groups:

1. 1st group will be control
2. 2nd group will take L-Arginine 500 mg.
3. 3rd group will undergo Tamsulosin 0.4 mg. I. Randomisation Randomization will be performed using computer generated random tables using stratified blocked randomization in 1:1:1 ratio.

Eligible patient will be informed on details of the study at our outpatient clinic. They also received written information.

Statistical Considerations And Data Analysis Sample size and statistical power The trial size was calculated concerning the primary endpoints by power calculations based on data from previous local comparative studies.

with an 80% power "beta", a 0.05 level of significance is considered "alpha" and with an expected 10% dropout rate.

ELIGIBILITY:
Inclusion criteria:

Patients older than 18 years old, ureter stones in size between 4 and 10 mm, single stone

Exclusion criteria:

Acute azotemia, stones larger than 10 mm, solitary kidney, symptomatic urinary system infection, impacted status, severe hydronephrosis, multiple or bilateral stones, pregnancy, anatomic urinary system abnormalities, benign prostate hyperplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Spontaneous stone expulsion rates (SER) | From 1st renal colic till the time of stone pass or for four weeks
  detect the rate at which stone pass from the ureter
Stone expulsion time | From 1st renal colic till the time of stone pass or for four weeks
  time at which stone pass
Number of daily colic episodes | number of colicky attack From 1st renal colic till the time of stone pass or for four weeks
  number of renal colic attack
Total required analgesic dosage | From 1st renal colic till the time of stone pass or for four weeks
  Total required analgesic dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
there are no need for this

REFERENCES:
- See also: most papper used — https://pubmed.ncbi.nlm.nih.gov/9008325/
- Available data/document: Study Protocol: ahmed-mahmoud@sohag.med.edu.eg — https://pubmed.ncbi.nlm.nih.gov/9008325/